CLINICAL TRIAL: NCT06467045
Title: Frequency of Adverse Events and Factors Causing Adverse Events in Pediatric Patients Receiving Sedation for Magnetic Resonance Imaging: Observational Study
Brief Title: Frequency of Adverse Events in Pediatric Patients Receiving Sedation for Magnetic Resonance Imaging
Status: Recruiting | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Kubra OZTURK, principal investigator, medical doctor, anesthesiology and reanimation, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: Sislietfal-kozturk-001
Record Dates: First submitted 2024-06-12; First posted 2024-06-20 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Sedation; Pediatric Anesthesia; Magnetic Resonance Imaging; Adverse Effect
Keywords: pediatric; adverse effects; magnetic resonance imaging; sedation; anesthesia
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients who received sedation for magnetic resonance imaging: All pediatric patients who received sedation for magnetic resonance imaging(MRI) in radiology unit will be added to this study. In the study, there is only one group. No comparisons are being made.
  Interventions: Other: Pediatric patients who received sedation for magnetic resonance imaging

INTERVENTIONS:
Other: Pediatric patients who received sedation for magnetic resonance imaging — Pediatric patients who underwent MRI under sedation will be prospectively observed. All non-intubated patients under the age of 16 will be included in the study. The demographic data, comorbidities, and medications of the patients, the procedures performed, the anesthetic drugs used, the expertise duration of the anesthesiologist, and the adverse effects encountered will be recorded.

SUMMARY:
Introduction:The application of anesthesia outside the operating room for pediatric patients has increased in recent years. For diagnostic and treatment follow-up purposes, magnetic resonance imaging (MRI) requires the pediatric patient to remain still, necessitating sedation. The study aimed to determine the frequency of adverse effects and influencing factors in pediatric patients undergoing sedation during MRI.

Methods: Between 19.06.2024 and 16.09.2024, estimated 500 pediatric patients who underwent MRI under sedation will be prospectively observed. All non-intubated patients under the age of 16 will be included in the study. The demographic data, comorbidities, and medications of the patients, the procedures performed, the anesthetic drugs used, the expertise duration of the anesthesiologist, and the adverse effects encountered will be recorded.

DETAILED DESCRIPTION:
In modern times, the application of anesthesia outside the operating room is increasingly common in pediatric patients for day procedures and imaging by clinics such as gastroenterology, cardiology, oncology, and radiology . In addition to the difficulty of airway control in pediatric patients, the risks increase in non-operating room settings due to the unfamiliarity of the environment and being far from the operating room. Moreover, anesthesia application is risky due to patient-independent reasons such as the insufficient number of auxiliary staff, the inadequate emergency experience of the personnel in the units, and the limited number and variety of materials . Therefore, anesthesia application in pediatric patients is specialized and requires an experienced anesthesia team .

MRI imaging is a noisy, long-lasting technique that must be performed motionless . Pediatric patients requiring MRI imaging often have congenital anomalies, accompanying diseases, and acquired diseases due to birth trauma. Additionally, the complication rate related to the procedure may increase with a cooperative, mobile child. For this reason, day procedures in pediatric patients should be performed under sedation .

Some of the undesirable side effects encountered after sedation in pediatric patients include nausea, vomiting, cough, laryngospasm, bronchospasm, pulmonary aspiration, allergic reactions, anaphylaxis, extravasation, neurological damage, cardiovascular instability, and cardiac arrest . Although serious side effects are rarely encountered, minor undesirable side effects are frequently encountered . Many studies emphasize that serious undesirable side effects following sedation and general anesthesia in children are respiratory complications .

In our country, pediatric anesthesia applications outside the operating room are performed in a limited number of centers. Although there are retrospective studies on pediatric patients undergoing magnetic resonance imaging under sedation in the literature, it has been observed that there is insufficient data on large-scale observational studies.

The hypothesis of the study is that the frequency of anesthesia-related adverse effects is high in pediatric patients sedated in non-operating room environments. The primary aim of our study is to determine the frequency of adverse events in pediatric patients sedated for magnetic resonance imaging. Secondly, the investigators aimed to identify the factors causing these adverse events.

ELIGIBILITY:
Inclusion Criteria:

* All non-intubated patients under the age of 16 were included in the study.

Exclusion Criteria:

* Intubated pediatric patients or older than 16 years patients were excluded.

Ages: 0 Days to 16 Years | Sex: All
Age Groups: Child
Study Population: 500 patients non-intubated under the age of 16 who underwent magnetic resonance imaging under sedation in the radiology unit will be included in the study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2024-09-21 (Estimated); Study Completion 2024-10-05 (Estimated)

PRIMARY OUTCOMES:
Perioperative adverse events | 1 hours
  In the study, the investigators will record the adverse effects includes respiratory, circulatory, neurological systems observed during the procedure. Respiratory adverse effects includes bronchospasm, laryngospasm, apnea, pulmonary aspiration, anaphylaxis. Circulatory system adverse affects includes hypotension, hypertension, cardiac arrest. In the study, neurological side effects such as glasgow coma scale impairment and convulsions will be recorded.
Postoperative adverse events | 2 hours
  In the study, the investigators will record the adverse effects includes respiratory, circulatory, neurological systems the 2 hours following the procedure. Respiratory adverse effects includes bronchospasm, laryngospasm, apnea, pulmonary aspiration, anaphylaxis. Circulatory system adverse affects includes hypotension, hypertension, cardiac arrest. In the study, neurological side effects such as glasgow coma scale impairment and convulsions will be recorded.

SECONDARY OUTCOMES:
Electrocardiography | 3 hours
  Participants will be monitored with electrocardiography during the procedure and 2 hours following it.
SPO2 | 3 hours
  Participants will be monitored with pulse oximetry during the procedure and 2 hours following it.
Caphnography | 3 hours
  Participants will be monitored with capnograph during the procedure and 2 hours following it.
Temperature Monitoring | 3 hours
  Participants will be monitored with temperature probe during the procedure and 2 hours following it.
Systolic and Diastolic blood pressure | 3 hours
  Participants will be monitored with blood pressure monitoring during the procedure and 2 hours following it.
Glasgow Coma Scale | 3 hours
  Participants will be followed with glaskow coma scale during the procedure and 2 hours following it. Minimum value is 3 and maximum value is 15.
Aldrete Score | 2 hours
  Participants will be assessed for recovery using the Aldrete score during the 2-hour follow-up period after the procedure. Minimum value is 0 and maximum value is 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Sisli Hamidiye Etfal Research and Training Hospital, Istanbul, Sarıyer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cosgrove P, Krauss BS, Cravero JP, Fleegler EW. Predictors of Laryngospasm During 276,832 Episodes of Pediatric Procedural Sedation. Ann Emerg Med. 2022 Dec;80(6):485-496. doi: 10.1016/j.annemergmed.2022.05.002. Epub 2022 Jun 23. PMID 35752522
- [Result] Habre W, Disma N, Virag K, Becke K, Hansen TG, Johr M, Leva B, Morton NS, Vermeulen PM, Zielinska M, Boda K, Veyckemans F; APRICOT Group of the European Society of Anaesthesiology Clinical Trial Network. Incidence of severe critical events in paediatric anaesthesia (APRICOT): a prospective multicentre observational study in 261 hospitals in Europe. Lancet Respir Med. 2017 May;5(5):412-425. doi: 10.1016/S2213-2600(17)30116-9. Epub 2017 Mar 28. PMID 28363725